CLINICAL TRIAL: NCT03357666
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Design, Multicenter Phase II Trial to Evaluate the Efficacy and Safety of HUDC_VT in Patients With Bacterial Vaginosis
Brief Title: Clinical Study to Evaluate the Efficacy of HUDC_VT in Patients With Bacterial Vaginosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haudongchun Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUDC-VT-201
Record Dates: First submitted 2017-11-23; First posted 2017-11-30 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Bacterial Vaginosis; HUDC_VT; Haudongchun
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Sodium Chloride; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- HUDC_VT(Glucose 200mg/Sodium chloride 200mg) (Experimental): Glucose 200mg/Sodium chloride 200mg, once a day, two tablets at a time for 7 days
  Interventions: Drug: HUDC_VT(Glucose 200mg/Sodium chloride 200mg)
- HUDC_VT(Glucose 400mg/Sodium chloride 200mg) (Experimental): Glucose 400mg/Sodium chloride 200mg, once a day, two tablets at a time for 7 days
  Interventions: Drug: HUDC_VT (Glucose 400mg/Sodium chloride 200mg)
- HUDC_VT(Glucose 400mg) (Experimental): Glucose 400mg, once a day, two tablets at a time for 7 days
  Interventions: Drug: HUDC_VT (Glucose 400mg)
- HUDC_VT(Sodium chloride 200mg) (Experimental): Sodium chloride 200mg, once a day, two tablets at a time for 7 days
  Interventions: Drug: HUDC_VT (Sodium chloride 200mg)
- Placebo (Placebo Comparator): Placebo, once a day, two tablets at a time for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HUDC_VT(Glucose 200mg/Sodium chloride 200mg) — Vaginal administration, two tablets once a day for 7 days
  Arms: HUDC_VT(Glucose 200mg/Sodium chloride 200mg)
Drug: HUDC_VT (Glucose 400mg/Sodium chloride 200mg) — Vaginal administration, two tablets once a day for 7 days
  Arms: HUDC_VT(Glucose 400mg/Sodium chloride 200mg)
Drug: HUDC_VT (Glucose 400mg) — Vaginal administration, two tablets once a day for 7 days
  Arms: HUDC_VT(Glucose 400mg)
Drug: HUDC_VT (Sodium chloride 200mg) — Vaginal administration, two tablets once a day for 7 days
  Arms: HUDC_VT(Sodium chloride 200mg)
Drug: Placebo — Vaginal administration, two tablets once a day for 7 days
  Arms: Placebo

SUMMARY:
The objective of the study is to confirm the pharmacological mechanism and evaluate the efficacy and safety after HUDC-VT administration compared to placebo in patients with bacterial vaginosis.

Vaginitis in adult women is extremely common and it often results in marked suffering. Epidemiologic studies indicate the high prevalence of vaginitis and the large number of causes in US.

The broad-spectrum antibiotics such as metronidazole have been used as a treatment of vaginitis.However, it is not desirable using of these antibiotics caused appearance of resistant bacterium and killing normal bacterium including lactobacillus.

In addition, it has been reported that long term treatment of antibiotics can be caused body toxicity through absolution by vagina.

The product, HUDC_VT, is a effective and safe vaginal tablet composed glucose and sodium chloride for treatment of vaginitis by preserving healthy condition in vagina.

ELIGIBILITY:
Inclusion Criteria:

1. Fertile women
2. Clinical diagnosis of bacterial vaginosis with criteria on below (3 out of 4 fulfilled criteria)

   * light gray adherent vaginal discharge
   * pH >4.5
   * Presence of clue cells ≥20%
   * Positive "10% KOH whiff test"
3. Nugent Score ≥ 4

Exclusion Criteria:

1. Pregnant or breast-feeding patient or planning pregnancy
2. Patient with candidiasis, Chlamydia trachomatis, Trichomonas vaginalis, Neisseria gonorrhoeae or Herpes simplex virus infection
3. Patient who received antifungal or antimicrobial therapy (systemic or intravaginal) within 30 days of randomization
4. Any condition or circumstance that would interfere with analysis of study results
5. Patient who have a plan to treat other disease (e.g cervical carcinoma) during clinical study period

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-03-22 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic cure rate of bacterial vaginosis at 2 weeks after last treatment | at 2 weeks after last treatment

SECONDARY OUTCOMES:
Therapeutic cure rate of bacterial vaginosis at last treatment | at 7 days
proportion of patients with Normal Nugent score | at 2 weeks after last treatment
proportion of patients with Normal Hay/Ison grade | at 2 weeks after last treatment
proportion of patients with Normal Vaginal Fluid pH | at 2 weeks after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: WonSeog Choi, Study Chair — Haudongchun Co., Ltd.
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No